CLINICAL TRIAL: NCT06541106
Title: Registry of Endovascular Treatment for Vertebrobasilar Dissecting Aneurysms in China
Acronym: VBDAs China
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University International Hospital (Other); The First People's Hospital of Lianyungang (Other); Chinese PLA General Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Yichang Central People's Hospital (Other); Taihe Hospital (Other); Liaocheng People's Hospital (Other); Binzhou People's Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Beijing Aerospace General Hospital (Other); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); The Second Hospital of Hebei Medical University (Other); Dalian Municipal Central Hospital (Other); Shijiazhuang Third Hospital (Unknown); Affiliated Hospital of Chengde Medical University (Other); Xingtai People's Hospital (Other); Taian City Central Hospital (Other); Wuhan Brain Hospital (Unknown)
Responsible Party: Principal Investigator, Ming Lv, MD, Beijing Tiantan Hospital
Other Study IDs: VBDAs China
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Dissecting Aneurysm of Cerebral Artery
Keywords: Vertebrobasilar dissecting aneurysms; Endovascular treatment; Prognosis; Hemorrhagic stroke
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conservative management group: Patients with unruptured VBDAs did not receive any interventional therapy (including endovascular therapy and microsurgery).
  Interventions: Other: Multi-disciplinary assessment
- Stent-assisted coiling group: Patients with unruptured VBDAs receive common stent and coils embolization.
- Flow diverter group: Patients with unruptured VBDAs receive flow diverter treatment.

INTERVENTIONS:
Other: Multi-disciplinary assessment — 1. Comprehensive evaluation was performed by multi-disciplinary experts to assess the prognosis of unruptured VBDAs and develop appropriate treatment strategies.
  2. Preoperative cranial MRI, CTA, DSA and other imaging tests were used to determine the aneurysm site, morphology, size, presence of compression symptoms, and whether it was accompanied by an intramural hematoma.
  Groups: Conservative management group

SUMMARY:
The incidence of vertebrobasilar dissecting aneurysms (VBDAs) is about 1/100,000~1.5/100,000, and it is one of the most important causes of stroke in young and middle-aged people. In recent years, with the development of medical imaging technology, the detection rate of this disease has been increasing year by year. The natural prognosis of VBDAs is complex and varied, with uncertainty: (1) it may have a benign course, and the imaging follow-up may show that the diseased vessels are repaired and improved or remain stable for a long period of time; (2) it may present with ischemic stroke caused by hemodynamic alteration or thromboembolism, which may result in severe neurological impairment; (3) it may occur as a result of rupture of aneurysms leading to subarachnoid hemorrhage, endangering the patient's life; (4) progressive enlargement of VBDAs causing occupying effects, which may be manifested as headache in mild cases, or hemiplegia of limbs and choking on drinking water in severe cases. Up to now, there is a lack of objective and uniform diagnostic and therapeutic guidelines for the natural regression of VBDAs and the benefits of surgery, and the treatment is mostly empirical, which makes it difficult to accurately determine the clinical prognosis of VBDAs and formulate appropriate treatment strategies.

Therefore, against the above background, we designed the present study. This study was a multicenter, prospective, registry study. We enrolled patients with unruptured VBDAs who met the inclusion and exclusion criteria, and a multi-disciplinary team formulated the treatment modalities for the patients, which were categorized into the conservative observation group, the stent-assisted coiling group, and the flow diverter group. The aim of our study was to investigate the effects of different treatment modalities on the prognosis of patients with VBDAs, as well as to stratify the risk factors of the patients, to explore the individualized treatment modalities of the patients, and to improve the diagnosis and treatment of this clinically refractory cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Patients diagnosis of "unruptured vertebrobasilar dissecting aneurysm".

Exclusion Criteria:

1. Patients did not undergo a cranial MRI;
2. Missing critical clinical baseline;
3. Missing pre-treatment imaging;
4. Receiving microsurgery;
5. The combination of other serious diseases during diagnosis will significantly affect the follow-up of patients;
6. CT/MRI shows intracranial hemorrhage or subarachnoid hemorrhage (SWI microbleeds are ignored).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosis of "unruptured vertebrobasilar dissecting aneurysm".
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Poor prognosis | 6 months, 1 year, 3 years, and 5 years after treatment.
  Defined as an mRS score of 3-6.
Aneurysm rupture | 6 months, 1 year, 3 years, and 5 years after treatment.
  Severe headache developed after treatment and was confirmed by CT as subarachnoid hemorrhage associated with VBDAs.

SECONDARY OUTCOMES:
Ischemic stroke | 6 months, 1 year, 3 years, and 5 years after treatment.
  Ischemic stroke refer to in-stent thrombosis, transient ischemic attack, or cerebral infarction associated with the treated vascular area.
Compression symptom | 6 months, 1 year, 3 years, and 5 years after treatment.
  Compression symptoms refer to cranial neuropathy or brainstem symptoms associated with aneurysm compression.
VBDA-related death | 6 months, 1 year, 3 years, and 5 years after treatment.
  Patients died during hospitalization or follow-up and were associated with VBDA. The causes of death were categorized as: aneurysm rupture, ischemic stroke, and compression symptoms.
Improvement of neurological dysfunction | 6 months, 1 year, 3 years, and 5 years after treatment.
  The modified Rankin score was used to evaluate neurological dysfunction: Grade 0, completely asymptomatic; Grade 1, able to complete all daily duties and activities despite symptoms, but without obvious dysfunction; Grade 2, mildly disabled, unable to complete all activities before illness, but does not need help, can take care of themself; Grade 3, moderately disabled, requires some help, but does not need help while walking; Grade 4, severely disabled, unable to walk independently, unable to meet their own needs without help from others; Grade 5, severely disabled, bedridden, incontinence, requiring continuous care And attention; Grade 6, death.
Rate of complete occlusion of aneurysms | 6 months, 1 year, 3 years, and 5 years after treatment.
  Complete occlusion of the aneurysm was confirmed by DSA, and then the rate of complete occlusion was compared between the groups.
Aneurysm recanalization | 6 months, 1 year, 3 years, and 5 years after treatment.
  Aneurysm recanalization was confirmed by DSA, and then the rate of aneurysm recanalization was compared between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Huang LT, Zhang M, Tong X. Cerebral revascularization for complex vertebrobasilar artery dissecting aneurysms. Neurosurg Rev. 2024 Apr 5;47(1):138. doi: 10.1007/s10143-024-02365-5. PMID 38578572
- [Background] Amoukhteh M, Hassankhani A, Valizadeh P, Jannatdoust P, Ghozy S, Kobeissi H, Kallmes DF. Flow diverters in the treatment of intracranial dissecting aneurysms: a systematic review and meta-analysis of safety and efficacy. J Neurointerv Surg. 2024 Sep 17;16(10):1005-1012. doi: 10.1136/jnis-2023-021117. PMID 38212103
- [Background] Dmytriw AA, Alrashed A, Enriquez-Marulanda A, Medhi G, Mendes Pereira V. Unruptured Intradural Posterior Circulation Dissecting/Fusiform Aneurysms Natural History and Treatment Outcome. Interv Neuroradiol. 2023 Feb;29(1):56-62. doi: 10.1177/15910199211068673. Epub 2021 Dec 22. PMID 34935531
- [Background] Nakatomi H, Kiyofuji S, Ono H, Tanaka M, Kamiyama H, Takizawa K, Imai H, Saito N, Shiokawa Y, Morita A, Flemming KD, Link MJ. Giant Fusiform and Dolichoectatic Aneurysms of the Basilar Trunk and Vertebrobasilar Junction-Clinicopathological and Surgical Outcome. Neurosurgery. 2020 Dec 15;88(1):82-95. doi: 10.1093/neuros/nyaa317. PMID 32745190
- [Background] Adeeb N, Ogilvy CS, Griessenauer CJ, Thomas AJ. Expanding the Indications for Flow Diversion: Treatment of Posterior Circulation Aneurysms. Neurosurgery. 2020 Jan 1;86(Suppl 1):S76-S84. doi: 10.1093/neuros/nyz344. PMID 31838535
- [Background] Cho DY, Kim BS, Choi JH, Park YK, Shin YS. The Fate of Unruptured Intracranial Vertebrobasilar Dissecting Aneurysm with Brain Stem Compression According to Different Treatment Modalities. AJNR Am J Neuroradiol. 2019 Nov;40(11):1924-1931. doi: 10.3174/ajnr.A6252. Epub 2019 Oct 10. PMID 31601577
- [Background] Frisoli FA, Srinivasan VM, Catapano JS, Rudy RF, Nguyen CL, Jonzzon S, Korson C, Karahalios K, Lawton MT. Vertebrobasilar dissecting aneurysms: microsurgical management in 42 patients. J Neurosurg. 2021 Dec 10;137(2):393-401. doi: 10.3171/2021.9.JNS21397. Print 2022 Aug 1. PMID 34891141
- [Background] Ahn SS, Kim BM, Suh SH, Kim DJ, Kim DI, Shin YS, Ha SY, Kwon YS. Spontaneous symptomatic intracranial vertebrobasilar dissection: initial and follow-up imaging findings. Radiology. 2012 Jul;264(1):196-202. doi: 10.1148/radiol.12112331. Epub 2012 May 1. PMID 22550310
- [Background] Zhang Y, Tian Z, Sui B, Wang Y, Liu J, Li M, Li Y, Jiang C, Yang X. Endovascular Treatment of Spontaneous Intracranial Fusiform and Dissecting Aneurysms: Outcomes Related to Imaging Classification of 309 Cases. World Neurosurg. 2017 Feb;98:444-455. doi: 10.1016/j.wneu.2016.11.074. Epub 2016 Nov 24. PMID 27890754
- [Background] Sonmez O, Brinjikji W, Murad MH, Lanzino G. Deconstructive and Reconstructive Techniques in Treatment of Vertebrobasilar Dissecting Aneurysms: A Systematic Review and Meta-Analysis. AJNR Am J Neuroradiol. 2015 Jul;36(7):1293-8. doi: 10.3174/ajnr.A4360. Epub 2015 May 7. PMID 25953763